CLINICAL TRIAL: NCT04802200
Title: Short-term Clinical Follow-up of the Vascular Closure Device MANTATM in Minimally Invasive Cardiac Surgery
Acronym: MANTA-MICS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: HAMDAN 2021
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Femoral Artery Injury; Aortic Valve Insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients operated from minimally invasive cardiac surgery: Patients operated between December 16, 2019 and june 30, 2021 from minimally invasive cardiac surgery with femoral cannulation for cardiopulmonary bypass in Dijon University hospital and in whom the MANTA device has been used for femoral artery closure
  Interventions: Other: Data collect

INTERVENTIONS:
Other: Data collect — Data collect following a vascular closure by MANTA

SUMMARY:
The percutaneous MANTA Vascular Closure Device is dedicated to the closure of large bore arteriotomies. It appears to be a safe and doable option for vascular access closure in patients undergoing transfemoral Transcatheter Aortic Valve Implantation. Data concerning safety and efficacy of MANTA Vascular Closure Device in Minimally Invasive Cardiac Surgery are scarce. This study aim to assess this novel collagen-based technology in minimal invasive aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agreeing to participate in the study
* Subject >= 18 years of age
* Patients operated between december 16, 2019 and june 30, 2021 from minimally invasive cardiac surgery with femoral cannulation for cardiopulmonary bypass in Dijon University Hospital
* Patients in whom the MANTA device has been used for femoral artery closure

Exclusion Criteria:

Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject adult voluntarily agreeing to participate in the study operated between December 16, 2019 and june 30, 2021 from minimally invasive cardiac surgery with femoral cannulation for cardiopulmonary bypass in Dijon University Hospital, in whom the MANTA device has been used for femoral artery closure
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Occurence of major access site vascular complications | 30 days
  according to the Valve Academic Research Consortium (VARC)-2 and Bleeding Academic Research Consortium (BARC)-2 definition criteria in postoperative period
Hemostasis success | 10 min
  Hemostasis at the puncture site of cutting the MANTA suture without need for manual or mechanical compression and without late re-bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France